CLINICAL TRIAL: NCT04813523
Title: Efficacy and Safety of Pembrolizumab Plus Neoadjuvant Chemotherapy With Cisplatin and 5-Fluorouracill Followed by Surgery in Patients With Locally Advanced Adenocarcinoma of Esophagogastric Junction
Brief Title: Pembrolizumab Plus Neoadjuvant Chemotherapy for Locally Advanced EGJ Adenocarcinoma
Acronym: KEYSTONE-003
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TianjinCIH20210169
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Adenocarcinoma of Esophagogastric Junction; Neoadjuvant Chemotherapy; Pembrolizumab
MeSH Terms: interventions — pembrolizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental: Pembrolizumab+Cisplatin+5-FU (Experimental): Participants receive preoperative pembrolizumab 200 mg intravenously (IV) every 3 weeks (Q3W), cisplatin 80 mg/m^2 IV Q3W, and 5-FU 600 mg/m^2/day IV infusion on Days 1 to 5. There are 3 cycels of preoprative therapy and 3 cycles of postoperative therapy.
  Interventions: Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Drug: Pembrolizumab Injection [Keytruda] — Neoadjuvant period: pembrolizumab 200mg IV, Q3W with three cycles. Adjuvant period: pembrolizumab 200 mg IV, Q3W, up to one year, which should be performed within 3-6 weeks after surgery.
  Other Names: Cisplatin; 5-FU

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of pembrolizumab plus cisplatin and 5-fluorouracil (5-FU) followed Surgery for locally advanced adenocarcinoma of esophagogastric junction

DETAILED DESCRIPTION:
The neoadjuvant chemotherapy/chemoradiotherapy with surgery is the standard treatment in NCCN guideline. But many patients refused or abandon radiotherapy because of the intolerable adverse effects. We designed a single-arm, open-label, phase II trial of pembrolizumab plus cisplatin and 5-fluorouracil (5-FU) followed by radical surgery for locally advanced adenocarcinoma of esophagogastric junction. The purpose of this study is to observe and evaluate the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed AEG, Siewert type I or II;
2. Potentially resectable cT3-4a, any N, M0 (AJCC 8 TNM classification);
3. Have a performance status of 0 or 1 on the ECOG Performance Scale;
4. Age 18-75 years old, both men and women;
5. Be willing and able to provide written informed consent/assent for the trial;
6. Demonstrate adequate organ function , all screening labs should be performed within 10 days of treatment initiation;
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
8. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. Newly-obtained is defined as a specimen obtained up to 4 weeks (28 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.

Exclusion Criteria:

1. Prior therapy (operation, radiotherapy, immunotherapy, or chemotherapy) for AEG;
2. Ineligibility or contraindication for esophagectomy;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug;
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs);
5. Has severe hypersensitivity and adverse events (≥Grade 3) to nivolumab and/or any PD-1/PD-L1 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response (MPR) | one month after surgery
  Viable tumor comprised ≤ 10% of resected tumor specimens

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  Time from the enrollment to disease relapse after complete resection or death from any cause
Overall survival (OS) | 24 months
  Time from the enrollment to death of any cause
Pathologic complete response (pCR) | one month after surgery
  No tumor residue of resected tumor specimens

CONTACTS AND LOCATIONS:
Locations (1):
- Department of minimally invasive esophageal surgery, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China